CLINICAL TRIAL: NCT00962780
Title: A Phase 3, Open-label, Single-Arm Trial to Evaluate the Safety, Tolerability and Immunogenicity of 2 and 3 Doses of 13vPnC in HIV-Infected Subjects 6 Years of Age and Older Who Have Not Been Previously Immunized With Pneumococcal Vaccine
Brief Title: Safety and Immunogenicity of 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) in HIV-Infected Subjects 6 Years of Age or Older Who Are Naive to Pneumococcal Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-3002; B1851021; NCT01098370 (obsolete NCT alias)
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: HIV Infections; Pneumococcal Infections
Keywords: vaccine; 13-valent pneumococcal conjugate vaccine; 23-valent pneumococcal polysaccharide vaccine; human immunodeficiency virus
MeSH Terms: conditions — HIV Infections; Pneumococcal Infections; Acquired Immunodeficiency Syndrome | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 3 doses of 13vPnC and 1 dose of 23vPS, each dose given approximately 1 month apart
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine (13vPnC); Biological: 23-valent Pneumococcal Polysaccharide Vaccine (23vPS); Procedure: Blood draw

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine (13vPnC) — 13vPnC; 3 vaccinations given at approximately 1 month intervals at visits 1-3
Biological: 23-valent Pneumococcal Polysaccharide Vaccine (23vPS) — 23vPS; 1 vaccination given at visit 4 (approximately 1 month after visit 3)
Procedure: Blood draw — Blood draw; 5 blood draws approximately 1 month apart taken prior to vaccination at visits 1-4 and visit 5 (approximately 1 month after visit 4).
Procedure: Blood draw — 1 or 2 blood draws for CD4+ T cell count and HIV viral load at least 6 weeks apart, if subject does not have 2 CD4+ T cell counts and HIV viral load counts within 6 months before visit 1.
  Other Names: Screening blood draw(s)

SUMMARY:
The study will evaluate the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate vaccine (13vPnC) in HIV-infected subjects 6 years of age or older who have not been previously immunized with a pneumococcal vaccine. All subjects will receive 3 doses of 13vPnC and 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS), with each dose given approximately 1 month apart.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus (HIV)-infected subjects aged 6 years or older
* Viral load < 50,000 copies/mL and CD4+ T cell count >= 200/uL within 6 months before study vaccination
* Receiving stable highly active antiretroviral therapy (HAART) or not currently receiving any antiretroviral therapy
* No previous vaccination with a pneumococcal vaccine
* Subject or parent/legal guardian able to complete an electronic diary

Exclusion Criteria:

* Acquired immune deficiency syndrome (AIDS) at time of enrollment
* Current illicit substance and/or alcohol abuse
* History of active chronic viral hepatitis
* Previous anaphylactic reaction to a vaccine or vaccine-related component
* Serious chronic disorders including metastatic malignancy and end-stage renal disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Romania (2):
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Constanța
- South Africa (7):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Soweto, Gauteng
  - Pfizer Investigational Site, Dundee, KwaZulu-Natal
  - Pfizer Investigational Site, Worcester, Western Cape
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Paarl

REFERENCES:
- [Derived] Bhorat AE, Madhi SA, Laudat F, Sundaraiyer V, Gurtman A, Jansen KU, Scott DA, Emini EA, Gruber WC, Schmoele-Thoma B. Immunogenicity and safety of the 13-valent pneumococcal conjugate vaccine in HIV-infected individuals naive to pneumococcal vaccination. AIDS. 2015 Jul 17;29(11):1345-54. doi: 10.1097/QAD.0000000000000689. PMID 25888646
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3002&StudyName=Safety%20and%20Immunogenicity%20of%2013-Valent%20pneumococcal%20conjugate%20vaccine%20%2813vPnC%29%20in%20HIV-Infected%20Subjects%206%20Years%20of%20Age%20or%20Older%20who

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC, 23vPS (Pediatric Participants): Participants older than or equal to [>=] 6 to less than [<] 18 years of age (pediatric participants) received 3 doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly 1 month apart, followed by 1 dose of 0.5 mL of 23-valent pneumococcal polysaccharide vaccine (23vPS) intramuscularly 1 month after 13vPnC Dose 3 (23vPS Dose).
- 13vPnC, 23vPS (Adult Participants): Participants >=18 years of age (adult participants) received 3 doses of 0.5 mL of 13vPnC intramuscularly 1 month apart, followed by 1 dose of 0.5 mL of 23vPS intramuscularly 1 month after 13vPnC Dose 3 (23vPS Dose).
Period: Overall Study
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants)
Started | 151 | 152
Vaccinated 13vPnC Dose 1 | 150 | 151
Vaccinated 13vPnC Dose 2 | 145 | 145
Vaccinated 13vPnC Dose 3 | 144 | 142
Vaccinated 23vPS Dose | 143 | 139
Completed | 141 | 138
Not Completed | 10 | 14
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 9 | 4
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | Total
Number analyzed (Participants) | 150 | 151 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (3.04) | 41.2 (8.45) | 25.8 (16.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 88 | 164
  Male | 74 | 63 | 137

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody From 1 Month After 13vPnC Dose 2 to 1 Month After 13vPnC Dose 3 in All Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month after 13vPnC Dose 2 to 1 month after 13vPnC Dose 3 were computed using the logarithmically transformed assay results. Confidence interval (CI) for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both 1 month after 13vPnC Dose 2 and after 13vPnC Dose 3 blood draws.
Time Frame: 1 month after 13vPnC Dose 2, 1 month after 13vPnC Dose 3
Population: Evaluable immunogenicity population:eligible participants who received vaccination as assigned;had blood drawn within pre-specified time-frames;had at least 1 valid, determinate assay result; had no major protocol violation. N (number of participants analyzed)=participants evaluable for this measure, n=participants evaluable for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Groups:
- 13vPnC, 23vPS (All Participants): Participants >=6 years of age (all participants) received 3 doses of 0.5 mL of 13vPnC intramuscularly 1 month apart, followed by 1 dose of 0.5 mL of 23vPS intramuscularly 1 month after 13vPnC Dose 3 (23vPS Dose).
Arm/Group | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 259
fold rise
  Serotype 1 (n = 248) | 1.03 [0.99 to 1.07]
  Serotype 3 (n = 238) | 1.05 [1.00 to 1.10]
  Serotype 4 (n = 257) | 1.09 [1.03 to 1.14]
  Serotype 5 (n = 257) | 1.01 [0.97 to 1.05]
  Serotype 6A (n = 249) | 1.02 [0.97 to 1.07]
  Serotype 6B (n = 257) | 1.04 [1.01 to 1.08]
  Serotype 7F (n = 259) | 1.10 [1.05 to 1.16]
  Serotype 9V (n = 259) | 1.05 [1.01 to 1.09]
  Serotype 14 (n = 259) | 1.04 [1.00 to 1.09]
  Serotype 18C (n = 259) | 0.99 [0.96 to 1.02]
  Serotype 19A (n = 259) | 0.99 [0.96 to 1.03]
  Serotype 19F (n = 252) | 1.06 [1.01 to 1.11]
  Serotype 23F (n = 258) | 1.09 [1.03 to 1.15]

2. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After 13vPnC Dose 3 Relative to 1 Month After 13vPnC Dose 2 in Pediatric, Adult and All Participants
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for pediatric, adult and all participants are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means were calculated using all participants with available data for both 1 month after 13vPnC Dose 2 and after 13vPnC Dose 3 blood draws. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after 13vPnC Dose 2, 1 month after 13vPnC Dose 3
Population: Evaluable immunogenicity population. Here "N" (number of participants analyzed) signifies all participants who were evaluable for this measure and "n" signifies all participants who were evaluable for specified serotype for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 128 | 131 | 259
microgram per milliliter (mcg/mL)
  Serotype 1: 13vPnC Dose 2 (n = 120, 128, 248) | 3.88 [3.30 to 4.57] | 3.95 [3.23 to 4.85] | 3.92 [3.44 to 4.46]
  Serotype 1: 13vPnC Dose 3 (n = 120, 128, 248) | 4.14 [3.56 to 4.83] | 3.92 [3.21 to 4.79] | 4.03 [3.55 to 4.57]
  Serotype 3: 13vPnC Dose 2 (n = 118, 120, 238) | 1.47 [1.25 to 1.74] | 0.97 [0.81 to 1.16] | 1.19 [1.05 to 1.35]
  Serotype 3: 13vPnC Dose 3 (n = 118, 120, 238) | 1.49 [1.26 to 1.76] | 1.06 [0.88 to 1.27] | 1.25 [1.11 to 1.42]
  Serotype 4: 13vPnC Dose 2 (n = 127, 130, 257) | 3.06 [2.54 to 3.69] | 2.97 [2.40 to 3.67] | 3.01 [2.62 to 3.47]
  Serotype 4: 13vPnC Dose 3 (n = 127, 130, 257) | 3.36 [2.84 to 3.97] | 3.19 [2.59 to 3.91] | 3.27 [2.87 to 3.73]
  Serotype 5: 13vPnC Dose 2 (n = 126, 131, 257) | 4.52 [3.78 to 5.39] | 5.77 [4.83 to 6.89] | 5.12 [4.51 to 5.80]
  Serotype 5: 13vPnC Dose 3 (n = 126, 131, 257) | 4.84 [4.12 to 5.70] | 5.53 [4.63 to 6.61] | 5.18 [4.60 to 5.85]
  Serotype 6A: 13vPnC Dose 2 (n = 119, 130, 249) | 7.66 [6.46 to 9.08] | 7.03 [5.71 to 8.67] | 7.33 [6.40 to 8.39]
  Serotype 6A: 13vPnC Dose 3 (n = 119, 130, 249) | 7.97 [6.81 to 9.33] | 7.04 [5.74 to 8.64] | 7.47 [6.56 to 8.51]
  Serotype 6B: 13vPnC Dose 2 (n = 127, 130, 257) | 11.43 [9.45 to 13.84] | 7.93 [6.51 to 9.65] | 9.50 [8.28 to 10.91]
  Serotype 6B: 13vPnC Dose 3 (n = 127, 130, 257) | 11.94 [10.01 to 14.24] | 8.28 [6.78 to 10.11] | 9.92 [8.67 to 11.35]
  Serotype 7F: 13vPnC Dose 2 (n = 128, 131, 259) | 4.25 [3.67 to 4.92] | 5.78 [4.81 to 6.95] | 4.96 [4.41 to 5.59]
  Serotype 7F: 13vPnC Dose 3 (n = 128, 131, 259) | 5.05 [4.38 to 5.82] | 5.90 [4.95 to 7.04] | 5.46 [4.88 to 6.12]
  Serotype 9V: 13vPnC Dose 2 (n = 128, 131, 259) | 4.81 [4.18 to 5.54] | 5.14 [4.27 to 6.19] | 4.98 [4.43 to 5.59]
  Serotype 9V: 13vPnC Dose 3 (n = 128, 131, 259) | 4.98 [4.35 to 5.70] | 5.48 [4.59 to 6.55] | 5.23 [4.67 to 5.84]
  Serotype 14: 13vPnC Dose 2 (n = 128, 131, 259) | 11.60 [8.76 to 15.35] | 15.14 [11.64 to 19.71] | 13.27 [10.96 to 16.08]
  Serotype 14: 13vPnC Dose 3 (n = 128, 131, 259) | 12.62 [9.75 to 16.33] | 15.13 [11.80 to 19.40] | 13.83 [11.57 to 16.53]
  Serotype 18C: 13vPnC Dose 2 (n = 128, 131, 259) | 3.79 [3.12 to 4.60] | 5.33 [4.34 to 6.54] | 4.50 [3.91 to 5.19]
  Serotype 18C: 13vPnC Dose 3 (n = 128, 131, 259) | 3.83 [3.19 to 4.60] | 5.18 [4.27 to 6.28] | 4.46 [3.90 to 5.10]
  Serotype 19A: 13vPnC Dose 2 (n = 128, 131, 259) | 14.38 [12.20 to 16.96] | 13.19 [11.06 to 15.75] | 13.77 [12.21 to 15.53]
  Serotype 19A: 13vPnC Dose 3 (n = 128, 131, 259) | 14.19 [12.17 to 16.54] | 13.18 [11.11 to 15.62] | 13.67 [12.20 to 15.32]
  Serotype 19F: 13vPnC Dose 2 (n = 124, 128, 252) | 5.78 [4.63 to 7.21] | 5.34 [4.17 to 6.84] | 5.55 [4.71 to 6.55]
  Serotype 19F: 13vPnC Dose 3 (n = 124, 128, 252) | 6.09 [4.98 to 7.44] | 5.67 [4.47 to 7.18] | 5.87 [5.03 to 6.85]
  Serotype 23F: 13vPnC Dose 2 (n = 127, 131, 258) | 6.45 [5.30 to 7.85] | 6.10 [4.86 to 7.66] | 6.27 [5.40 to 7.28]
  Serotype 23F: 13vPnC Dose 3 (n = 127, 131, 258) | 6.64 [5.55 to 7.94] | 7.06 [5.65 to 8.82] | 6.85 [5.94 to 7.90]

3. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) 1 Month After 13vPnC Dose 3 Relative to 1 Month After 13vPnC Dose 2 in Pediatric, Adult and All Participants
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of pediatric, adult and all participants using a microcolony OPA (mcOPA) assay. GMT (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for both 1 month after 13vPnC Dose 2 and after 13vPnC Dose 3 blood draws. CI for GMT were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after 13vPnC Dose 2, 1 month after 13vPnC Dose 3
Population: Evaluable immunogenicity population. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants with valid and determinate assay results for specified serotype at both 1 month after 13vPnC Dose 2 and after 13vPnC Dose 3 blood draws for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 127 | 129 | 256
titers
  Serotype 1: 13vPnC Dose 2 (n = 126, 127, 253) | 51 [37.2 to 70.0] | 54 [38.7 to 74.2] | 52 [41.8 to 65.5]
  Serotype 1: 13vPnC Dose 3 (n = 126, 127, 253) | 69 [51.6 to 91.4] | 69 [51.3 to 92.0] | 69 [56.1 to 84.1]
  Serotype 3: 13vPnC Dose 2 (n = 127, 129, 256) | 81 [64.1 to 102.0] | 48 [37.9 to 61.5] | 62 [52.6 to 73.9]
  Serotype 3: 13vPnC Dose 3 (n = 127, 129, 256) | 114 [94.5 to 137.8] | 79 [62.1 to 99.9] | 95 [81.3 to 110.3]
  Serotype 4: 13vPnC Dose 2 (n = 117, 126, 243) | 2509 [1922.3 to 3274.2] | 1620 [1211.2 to 2167.4] | 2000 [1639.8 to 2439.1]
  Serotype 4: 13vPnC Dose 3 (n = 117, 126, 243) | 3246 [2697.1 to 3906.3] | 1944 [1465.3 to 2579.7] | 2488 [2092.1 to 2959.8]
  Serotype 5: 13vPnC Dose 2 (n = 122, 124, 246) | 159 [109.2 to 232.2] | 104 [69.1 to 156.9] | 129 [97.3 to 169.7]
  Serotype 5: 13vPnC Dose 3 (n = 122, 124, 246) | 267 [191.3 to 371.5] | 142 [97.5 to 206.7] | 194 [150.8 to 249.7]
  Serotype 6A: 13vPnC Dose 2 (n = 125, 124, 249) | 5560 [4378.4 to 7060.9] | 2425 [1790.7 to 3284.5] | 3678 [3016.2 to 4485.6]
  Serotype 6A: 13vPnC Dose 3 (n = 125, 124, 249) | 7758 [6314.2 to 9531.2] | 3239 [2488.5 to 4215.9] | 5022 [4216.8 to 5979.9]
  Serotype 6B: 13vPnC Dose 2 (n = 121, 128, 249) | 5449 [4365.1 to 6801.1] | 2724 [2004.8 to 3701.0] | 3815 [3140.9 to 4634.1]
  Serotype 6B: 13vPnC Dose 3 (n = 121, 128, 249) | 7151 [5828.2 to 8773.9] | 3723 [2771.1 to 5002.5] | 5113 [4250.1 to 6150.5]
  Serotype 7F: 13vPnC Dose 2 (n = 125, 127, 252) | 3494 [2772.8 to 4403.3] | 2255 [1739.6 to 2923.6] | 2802 [2352.6 to 3338.0]
  Serotype 7F: 13vPnC Dose 3 (n = 125, 127, 252) | 4638 [3889.7 to 5529.4] | 2702 [2130.3 to 3428.2] | 3533 [3037.4 to 4108.5]
  Serotype 9V: 13vPnC Dose 2 (n = 118, 127, 245) | 3339 [2461.4 to 4530.3] | 1432 [998.6 to 2054.9] | 2153 [1690.3 to 2743.3]
  Serotype 9V: 13vPnC Dose 3 (n = 118, 127, 245) | 4714 [3731.5 to 5955.4] | 2004 [1416.5 to 2836.1] | 3026 [2434.3 to 3761.4]
  Serotype 14: 13vPnC Dose 2 (n = 117, 127, 244) | 3704 [2906.5 to 4719.5] | 1342 [1010.1 to 1782.1] | 2183 [1792.2 to 2659.6]
  Serotype 14: 13vPnC Dose 3 (n = 117, 127, 244) | 3963 [3195.8 to 4914.2] | 1480 [1150.3 to 1903.9] | 2373 [1988.4 to 2832.8]
  Serotype 18C: 13vPnC Dose 2 (n = 117, 121, 238) | 4635 [3609.7 to 5951.8] | 1349 [947.0 to 1921.5] | 2475 [1965.7 to 3115.4]
  Serotype 18C: 13vPnC Dose 3 (n = 117, 121, 238) | 5579 [4423.7 to 7036.9] | 1787 [1272.8 to 2508.5] | 3127 [2515.2 to 3888.6]
  Serotype 19A: 13vPnC Dose 2 (n = 125, 127, 252) | 684 [519.2 to 902.1] | 458 [332.5 to 631.2] | 559 [452.3 to 690.9]
  Serotype 19A: 13vPnC Dose 3 (n = 125, 127, 252) | 1002 [814.5 to 1232.3] | 613 [465.6 to 806.4] | 782 [657.2 to 930.5]
  Serotype 19F: 13vPnC Dose 2 (n = 122, 118, 240) | 717 [495.6 to 1036.7] | 315 [196.7 to 506.0] | 479 [354.4 to 646.9]
  Serotype 19F: 13vPnC Dose 3 (n = 122, 118, 240) | 1152 [864.2 to 1535.0] | 597 [397.9 to 897.1] | 834 [650.1 to 1070.2]
  Serotype 23F: 13vPnC Dose 2 (n = 120, 126, 246) | 1477 [1086.2 to 2008.2] | 409 [271.9 to 614.0] | 765 [585.2 to 999.4]
  Serotype 23F: 13vPnC Dose 3 (n = 120, 126, 246) | 2327 [1844.2 to 2935.9] | 671 [449.8 to 1000.3] | 1231 [963.0 to 1572.5]

4. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) From 1 Month After 13vPnC Dose 2 to 1 Month After 13vPnC Dose 3 in Pediatric, Adult and All Participants
Description: as for outcome 1
Time Frame: 1 month after 13vPnC Dose 2, 1 month after 13vPnC Dose 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 127 | 129 | 256
fold rise
  Serotype 1 (n = 126, 127, 253) | 1.3 [1.13 to 1.61] | 1.3 [1.09 to 1.51] | 1.3 [1.16 to 1.48]
  Serotype 3 (n = 127, 129, 256) | 1.4 [1.25 to 1.59] | 1.6 [1.45 to 1.83] | 1.5 [1.40 to 1.65]
  Serotype 4 (n = 117, 126, 243) | 1.3 [1.10 to 1.52] | 1.2 [1.07 to 1.34] | 1.2 [1.13 to 1.37]
  Serotype 5 (n = 122, 124, 246) | 1.7 [1.36 to 2.06] | 1.4 [1.17 to 1.59] | 1.5 [1.33 to 1.72]
  Serotype 6A (n = 125, 124, 249) | 1.4 [1.22 to 1.60] | 1.3 [1.15 to 1.55] | 1.4 [1.23 to 1.51]
  Serotype 6B (n = 121, 128, 249) | 1.3 [1.18 to 1.46] | 1.4 [1.20 to 1.56] | 1.3 [1.23 to 1.46]
  Serotype 7F (n = 125, 127, 252) | 1.3 [1.15 to 1.53] | 1.2 [1.03 to 1.40] | 1.3 [1.14 to 1.40]
  Serotype 9V (n = 118, 127, 245) | 1.4 [1.16 to 1.72] | 1.4 [1.18 to 1.65] | 1.4 [1.24 to 1.60]
  Serotype 14 (n = 117, 127, 244) | 1.1 [0.95 to 1.20] | 1.1 [0.98 to 1.24] | 1.1 [1.00 to 1.18]
  Serotype 18C (n = 117, 121, 238) | 1.2 [1.10 to 1.32] | 1.3 [1.08 to 1.63] | 1.3 [1.13 to 1.42]
  Serotype 19A (n = 125, 127, 252) | 1.5 [1.27 to 1.68] | 1.3 [1.18 to 1.52] | 1.4 [1.27 to 1.54]
  Serotype 19F (n = 122, 118, 240) | 1.6 [1.31 to 1.97] | 1.9 [1.45 to 2.48] | 1.7 [1.48 to 2.06]
  Serotype 23F (n = 120, 126, 246) | 1.6 [1.31 to 1.90] | 1.6 [1.34 to 2.02] | 1.6 [1.40 to 1.85]

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody From 1 Month After 13vPnC Dose 2 to 1 Month After 13vPnC Dose 3 in Pediatric and Adult Participants
Description: as for outcome 1
Time Frame: 1 month after 13vPnC Dose 2, 1 month after 13vPnC Dose 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants)
Number analyzed (Participants) | 128 | 131
fold rise
  Serotype 1 (n = 120, 128) | 1.07 [1.01 to 1.13] | 0.99 [0.93 to 1.06]
  Serotype 3 (n = 118, 120) | 1.01 [0.95 to 1.08] | 1.09 [1.02 to 1.16]
  Serotype 4 (n = 127, 130) | 1.10 [1.02 to 1.18] | 1.07 [1.00 to 1.16]
  Serotype 5 (n = 126, 131) | 1.07 [1.01 to 1.14] | 0.96 [0.91 to 1.01]
  Serotype 6A (n = 119, 130) | 1.04 [0.96 to 1.12] | 1.00 [0.95 to 1.06]
  Serotype 6B (n = 127, 130) | 1.04 [0.99 to 1.10] | 1.04 [0.99 to 1.11]
  Serotype 7F (n = 128, 131) | 1.19 [1.12 to 1.27] | 1.02 [0.95 to 1.10]
  Serotype 9V (n = 128, 131) | 1.03 [0.98 to 1.09] | 1.07 [1.02 to 1.12]
  Serotype 14 (n = 128, 131) | 1.09 [1.02 to 1.16] | 1.00 [0.95 to 1.05]
  Serotype 18C (n = 128, 131) | 1.01 [0.96 to 1.07] | 0.97 [0.93 to 1.01]
  Serotype 19A (n = 128, 131) | 0.99 [0.93 to 1.04] | 1.00 [0.96 to 1.04]
  Serotype 19F (n = 124, 128) | 1.05 [0.98 to 1.13] | 1.06 [0.99 to 1.14]
  Serotype 23F (n = 127, 131) | 1.03 [0.96 to 1.11] | 1.16 [1.07 to 1.26]

6. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody Before and 1 Month After 13vPnC Dose 1 in Pediatric, Adult and All Participants
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for pediatric, adult and all participants are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for both the before and after 13vPnC Dose 1 blood draws. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1
Population: Evaluable immunogenicity population. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants with valid and determinate assay results for specified serotype at both the before and 1 month after 13vPnC Dose 1 blood draws for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 133 | 137 | 270
mcg/mL
  Serotype 1: Before 13vPnC Dose 1 (n=78,122,200) | 1.03 [0.72 to 1.48] | 0.82 [0.63 to 1.06] | 0.90 [0.73 to 1.10]
  Serotype 1: After 13vPnC Dose 1 (n=78,122,200) | 3.78 [2.97 to 4.80] | 4.00 [3.19 to 5.01] | 3.91 [3.32 to 4.61]
  Serotype 3: Before 13vPnC Dose 1 (n=99,127,226) | 0.83 [0.62 to 1.11] | 0.47 [0.37 to 0.58] | 0.60 [0.50 to 0.72]
  Serotype 3: After 13vPnC Dose 1 (n=99,127,226) | 1.25 [0.99 to 1.58] | 0.75 [0.62 to 0.92] | 0.94 [0.81 to 1.09]
  Serotype 4: Before 13vPnC Dose 1 (n=95,127,222) | 0.19 [0.14 to 0.25] | 0.35 [0.28 to 0.45] | 0.27 [0.22 to 0.33]
  Serotype 4: After 13vPnC Dose 1 (n=95,127,222) | 2.62 [1.97 to 3.50] | 2.91 [2.26 to 3.75] | 2.79 [2.31 to 3.36]
  Serotype 5: Before 13vPnC Dose 1 (n=122,137,259) | 4.18 [3.42 to 5.12] | 3.38 [2.84 to 4.02] | 3.74 [3.28 to 4.27]
  Serotype 5: After 13vPnC Dose 1 (n=122,137,259) | 4.81 [3.98 to 5.80] | 5.53 [4.63 to 6.61] | 5.18 [4.55 to 5.89]
  Serotype 6A: Before 13vPnC Dose 1 (n=99,136,235) | 6.22 [5.19 to 7.45] | 2.67 [2.24 to 3.18] | 3.81 [3.32 to 4.37]
  Serotype 6A: After 13vPnC Dose 1 (n=99,136,235) | 7.31 [6.07 to 8.79] | 6.77 [5.38 to 8.51] | 6.99 [6.00 to 8.15]
  Serotype 6B: Before 13vPnC Dose 1 (n=131,134,265) | 5.52 [4.59 to 6.64] | 3.23 [2.69 to 3.88] | 4.21 [3.69 to 4.81]
  Serotype 6B: After 13vPnC Dose 1 (n=131,134,265) | 10.26 [8.37 to 12.58] | 7.29 [5.81 to 9.15] | 8.63 [7.41 to 10.06]
  Serotype 7F: Before 13vPnC Dose 1 (n=111,134,245) | 0.85 [0.63 to 1.14] | 1.14 [0.94 to 1.37] | 1.00 [0.84 to 1.18]
  Serotype 7F: After 13vPnC Dose 1 (n=111,134,245) | 4.34 [3.68 to 5.11] | 5.57 [4.57 to 6.78] | 4.97 [4.36 to 5.67]
  Serotype 9V: Before 13vPnC Dose 1 (n=129,137,266) | 2.10 [1.74 to 2.54] | 1.56 [1.30 to 1.86] | 1.80 [1.58 to 2.05]
  Serotype 9V: After 13vPnC Dose 1 (n=129,137,266) | 4.77 [4.08 to 5.57] | 5.16 [4.24 to 6.27] | 4.97 [4.38 to 5.63]
  Serotype 14: Before 13vPnC Dose 1 (n=113,136,249) | 0.76 [0.57 to 1.03] | 2.45 [1.94 to 3.09] | 1.44 [1.18 to 1.76]
  Serotype 14: After 13vPnC Dose 1 (n=113,136,249) | 12.04 [8.48 to 17.10] | 16.46 [12.38 to 21.90] | 14.28 [11.44 to 17.84]
  Serotype 18C: Before 13vPnC Dose 1 (n=127,134,261) | 0.66 [0.52 to 0.85] | 0.85 [0.69 to 1.04] | 0.75 [0.64 to 0.88]
  Serotype 18C: After 13vPnC Dose 1 (n=127,134,261) | 3.92 [3.14 to 4.91] | 5.55 [4.51 to 6.84] | 4.69 [4.02 to 5.46]
  Serotype 19A: Before 13vPnC Dose 1 (n=133,137,270) | 7.51 [6.34 to 8.90] | 4.78 [4.04 to 5.66] | 5.97 [5.29 to 6.74]
  Serotype 19A: After 13vPnC Dose 1 (n=133,137,270) | 13.28 [11.11 to 15.87] | 13.03 [10.75 to 15.80] | 13.15 [11.54 to 14.99]
  Serotype 19F: Before 13vPnC Dose 1 (n=93,126,219) | 1.36 [1.06 to 1.75] | 1.36 [1.07 to 1.73] | 1.36 [1.14 to 1.62]
  Serotype 19F: After 13vPnC Dose 1 (n=93,126,219) | 4.62 [3.55 to 6.02] | 4.98 [3.74 to 6.62] | 4.82 [3.96 to 5.88]
  Serotype 23F: Before 13vPnC Dose 1 (n=126,137,263) | 2.29 [1.83 to 2.86] | 1.61 [1.31 to 1.96] | 1.90 [1.64 to 2.21]
  Serotype 23F: After 13vPnC Dose 1 (n=126,137,263) | 5.65 [4.66 to 6.86] | 5.30 [4.16 to 6.75] | 5.47 [4.68 to 6.39]

7. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody From Before 13vPnC Dose 1 to 1 Month After 13vPnC Dose 1 in Pediatric, Adult and All Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC Dose 1 to 1 month after 13vPnC Dose 1 were computed using the logarithmically transformed assay results. Confidence interval (CI) for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before 13vPnC Dose and after 13vPnC Dose 1 blood draws.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 133 | 137 | 270
fold rise
  Serotype 1 (n = 78, 122, 200) | 3.67 [2.70 to 4.99] | 4.88 [3.87 to 6.15] | 4.37 [3.63 to 5.25]
  Serotype 3 (n = 99, 127, 226) | 1.51 [1.27 to 1.79] | 1.62 [1.43 to 1.83] | 1.57 [1.42 to 1.74]
  Serotype 4 (n = 95, 127, 222) | 14.02 [10.55 to 18.62] | 8.29 [6.55 to 10.49] | 10.38 [8.64 to 12.47]
  Serotype 5 (n = 122, 137, 259) | 1.15 [1.06 to 1.25] | 1.64 [1.44 to 1.85] | 1.38 [1.28 to 1.50]
  Serotype 6A (n = 99, 136, 235) | 1.18 [1.02 to 1.35] | 2.54 [2.09 to 3.07] | 1.83 [1.60 to 2.10]
  Serotype 6B (n = 131, 134, 265) | 1.86 [1.55 to 2.22] | 2.26 [1.87 to 2.72] | 2.05 [1.80 to 2.33]
  Serotype 7F (n = 111, 134, 245) | 5.11 [3.92 to 6.65] | 4.90 [3.99 to 6.03] | 4.99 [4.24 to 5.88]
  Serotype 9V (n = 129, 137, 266) | 2.27 [1.97 to 2.61] | 3.32 [2.76 to 3.99] | 2.76 [2.45 to 3.10]
  Serotype 14 (n = 113, 136, 249) | 15.79 [11.84 to 21.05] | 6.73 [5.17 to 8.76] | 9.91 [8.11 to 12.11]
  Serotype 18C (n = 127, 134, 261) | 5.92 [4.64 to 7.55] | 6.55 [5.23 to 8.20] | 6.23 [5.29 to 7.35]
  Serotype 19A (n = 133, 137, 270) | 1.77 [1.55 to 2.02] | 2.73 [2.31 to 3.21] | 2.20 [1.98 to 2.45]
  Serotype 19F (n = 93, 126, 219) | 3.39 [2.71 to 4.25] | 3.66 [2.96 to 4.52] | 3.54 [3.04 to 4.13]
  Serotype 23F (n = 126, 137, 263) | 2.47 [2.02 to 3.02] | 3.30 [2.71 to 4.03] | 2.87 [2.49 to 3.31]

8. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) Before and 1 Month After 13vPnC Dose 1 in Pediatric, Adult and All Participants
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of pediatric, adult and all participants using a microcolony OPA (mcOPA) assay. GMT (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for both the before and after 13vPnC Dose 1 blood draws. CI for GMT were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 129 | 128 | 257
titers
  Serotype 1: Before 13vPnC Dose 1 (n=129,127,256) | 5 [4.3 to 5.8] | 5 [4.3 to 5.2] | 5 [4.4 to 5.3]
  Serotype 1: After 13vPnC Dose 1 (n=129,127,256) | 49 [35.3 to 68.1] | 57 [41.6 to 79.3] | 53 [42.2 to 66.7]
  Serotype 3: Before 13vPnC Dose 1 (n=126,128,254) | 8 [6.6 to 10.8] | 5 [4.5 to 5.8] | 7 [5.7 to 7.5]
  Serotype 3: After 13vPnC Dose 1 (n=126,128,254) | 41 [31.7 to 52.6] | 21 [16.3 to 27.1] | 29 [24.3 to 35.1]
  Serotype 4: Before 13vPnC Dose 1 (n=108,119,227) | 25 [15.2 to 41.7] | 27 [17.0 to 42.1] | 26 [18.6 to 36.3]
  Serotype 4: After 13vPnC Dose 1 (n=108,119,227) | 2247 [1611.9 to 3131.4] | 1372 [958.8 to 1963.7] | 1735 [1356.9 to 2218.3]
  Serotype 5: Before 13vPnC Dose 1 (n=125,122,247) | 5 [4.5 to 6.7] | 6 [4.8 to 6.8] | 6 [4.9 to 6.4]
  Serotype 5: After 13vPnC Dose 1 (n=125,122,247) | 79 [52.5 to 118.0] | 123 [81.8 to 186.3] | 98 [73.7 to 131.1]
  Serotype 6A: Before 13vPnC Dose 1 (n=99,98,197) | 157 [84.4 to 292.5] | 61 [35.1 to 106.8] | 98 [64.6 to 149.4]
  Serotype 6A: After 13vPnC Dose 1 (n=99,98,197) | 3480 [2460.1 to 4921.8] | 1543 [984.4 to 2418.5] | 2322 [1743.1 to 3092.9]
  Serotype 6B: Before 13vPnC Dose 1 (n=101,120,221) | 279 [155.5 to 501.1] | 231 [143.4 to 372.5] | 252 [174.1 to 364.6]
  Serotype 6B: After 13vPnC Dose 1 (n=101,120,221) | 3852 [2888.3 to 5137.8] | 2099 [1455.6 to 3028.2] | 2771 [2179.2 to 3522.5]
  Serotype 7F: Before 13vPnC Dose 1 (n=110,113,223) | 416 [253.5 to 682.9] | 38 [22.9 to 64.6] | 124 [84.3 to 183.8]
  Serotype 7F: After 13vPnC Dose 1 (n=110,113,223) | 3775 [3019.4 to 4720.1] | 2005 [1443.9 to 2783.1] | 2739 [2237.5 to 3353.5]
  Serotype 9V: Before 13vPnC Dose 1 (n=109,117,226) | 152 [87.2 to 266.2] | 69 [40.7 to 117.2] | 101 [68.8 to 148.6]
  Serotype 9V: After 13vPnC Dose 1 (n=109,117,226) | 2533 [1822.7 to 3520.3] | 1231 [836.1 to 1812.2] | 1743 [1347.0 to 2256.4]
  Serotype 14: Before 13vPnC Dose 1 (n=107,126,233) | 328 [201.4 to 535.5] | 123 [79.6 to 191.4] | 193 [139.0 to 269.2]
  Serotype 14: After 13vPnC Dose 1 (n=107,126,233) | 3571 [2772.2 to 4600.1] | 1277 [944.9 to 1725.8] | 2048 [1660.8 to 2524.9]
  Serotype 18C: Before 13vPnC Dose 1 (n=95,120,215) | 42 [21.9 to 79.0] | 25 [15.5 to 39.6] | 31 [21.2 to 45.8]
  Serotype 18C: After 13vPnC Dose 1 (n=95,120,215) | 2821 [1891.1 to 4208.9] | 1031 [671.3 to 1584.6] | 1609 [1188.2 to 2178.5]
  Serotype 19A: Before 13vPnC Dose 1 (n=129,128,257) | 28 [19.1 to 40.8] | 23 [16.7 to 32.7] | 26 [19.9 to 32.9]
  Serotype 19A: After 13vPnC Dose 1 (n=129,128,257) | 506 [381.9 to 671.7] | 390 [275.2 to 552.8] | 445 [355.7 to 555.9]
  Serotype 19F: Before 13vPnC Dose 1 (n=123,123,246) | 11 [7.6 to 15.5] | 14 [9.5 to 20.1] | 12 [9.5 to 15.8]
  Serotype 19F: After 13vPnC Dose 1 (n=123,123,246) | 425 [285.3 to 632.5] | 214 [130.4 to 352.3] | 302 [219.3 to 415.2]
  Serotype 23F: Before 13vPnC Dose 1 (n=118,125,243) | 14 [9.3 to 22.0] | 7 [5.3 to 9.0] | 10 [7.6 to 12.7]
  Serotype 23F: After 13vPnC Dose 1 (n=118,125,243) | 587 [379.3 to 907.7] | 140 [86.6 to 227.6] | 281 [200.8 to 393.7]

9. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) From Before 13vPnC Dose 1 to 1 Month After 13vPnC Dose 1 in Pediatric, Adult and All Participants
Description: as for outcome 7
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 129 | 128 | 257
fold rise
  Serotype 1 (n = 129, 127, 256) | 9.8 [6.97 to 13.81] | 12.2 [8.84 to 16.84] | 10.9 [8.65 to 13.81]
  Serotype 3 (n = 126, 128, 254) | 4.8 [3.72 to 6.30] | 4.1 [3.22 to 5.30] | 4.5 [3.73 to 5.35]
  Serotype 4 (n = 108, 119, 227) | 89.4 [51.43 to 155.31] | 51.3 [31.16 to 84.59] | 66.8 [46.17 to 96.75]
  Serotype 5 (n = 125, 122, 247) | 14.4 [9.56 to 21.67] | 21.7 [14.55 to 32.32] | 17.6 [13.25 to 23.44]
  Serotype 6A (n = 99, 98, 197) | 22.2 [12.61 to 38.90] | 25.2 [14.51 to 43.83] | 23.6 [15.98 to 34.94]
  Serotype 6B (n = 101, 120, 221) | 13.8 [8.12 to 23.45] | 9.1 [5.91 to 13.95] | 11.0 [7.87 to 15.37]
  Serotype 7F (n = 110, 113, 223) | 9.1 [5.79 to 14.23] | 52.2 [31.42 to 86.57] | 22.0 [15.42 to 31.42]
  Serotype 9V (n = 109, 117, 226) | 16.6 [9.71 to 28.47] | 17.8 [10.53 to 30.18] | 17.2 [11.87 to 25.04]
  Serotype 14 (n = 107, 126, 233) | 10.9 [6.79 to 17.41] | 10.3 [6.82 to 15.70] | 10.6 [7.76 to 14.44]
  Serotype 18C (n = 95, 120, 215) | 67.9 [35.25 to 130.73] | 41.6 [24.59 to 70.26] | 51.6 [34.27 to 77.78]
  Serotype 19A (n = 129, 128, 257) | 18.1 [12.52 to 26.25] | 16.7 [11.78 to 23.61] | 17.4 [13.51 to 22.38]
  Serotype 19F (n = 123, 123, 246) | 39.0 [24.56 to 62.05] | 15.5 [9.77 to 24.65] | 24.6 [17.69 to 34.25]
  Serotype 23F (n = 118, 125, 243) | 41.1 [24.94 to 67.81] | 20.2 [12.78 to 32.05] | 28.6 [20.34 to 40.10]

10. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After 13vPnC Dose 3 and 1 Month After 23vPS Dose in Pediatric, Adult and All Participants
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for pediatric, adult and all participants are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for both after 13vPnC Dose 3 and after 23vPS Dose blood draws. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after 13vPnC Dose 3, 1 month after 23vPS Dose
Population: Evaluable immunogenicity population. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants with valid and determinate assay results for specified serotype at both 1 month after 13vPnC Dose 3 and after 23vPS Dose blood draws for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 133 | 130 | 263
mcg/mL
  Serotype 1: After 13vPnC Dose 3 (n=128,127,255) | 4.08 [3.53 to 4.73] | 3.94 [3.22 to 4.82] | 4.01 [3.54 to 4.54]
  Serotype 1: After 23vPS Dose (n=128,127,255) | 4.42 [3.80 to 5.14] | 4.02 [3.32 to 4.85] | 4.21 [3.74 to 4.75]
  Serotype 3: After 13vPnC Dose 3 (n=124,118,242) | 1.49 [1.27 to 1.75] | 1.04 [0.87 to 1.26] | 1.25 [1.11 to 1.42]
  Serotype 3: After 23vPS Dose (n=124,118,242) | 1.65 [1.42 to 1.92] | 0.98 [0.82 to 1.17] | 1.28 [1.14 to 1.44]
  Serotype 4: After 13vPnC Dose 3 (n=133,128,261) | 3.29 [2.79 to 3.87] | 3.19 [2.59 to 3.93] | 3.24 [2.84 to 3.70]
  Serotype 4: After 23vPS Dose (n=133,128,261) | 3.28 [2.77 to 3.88] | 3.01 [2.44 to 3.72] | 3.15 [2.75 to 3.59]
  Serotype 5: After 13vPnC Dose 3 (n=132,130,262) | 4.73 [4.02 to 5.57] | 5.54 [4.64 to 6.63] | 5.12 [4.54 to 5.78]
  Serotype 5: After 23vPS Dose (n=132,130,262) | 5.08 [4.33 to 5.95] | 6.20 [5.23 to 7.35] | 5.61 [4.99 to 6.30]
  Serotype 6A: After 13vPnC Dose 3 (n=122,129,251) | 8.20 [6.99 to 9.61] | 7.07 [5.75 to 8.69] | 7.60 [6.67 to 8.66]
  Serotype 6A: After 23vPS Dose (n=122,129,251) | 7.98 [6.85 to 9.31] | 6.71 [5.51 to 8.17] | 7.30 [6.44 to 8.27]
  Serotype 6B: After 13vPnC Dose 3 (n=133,129,262) | 12.25 [10.31 to 14.55] | 8.29 [6.78 to 10.13] | 10.10 [8.84 to 11.55]
  Serotype 6B: After 23vPS Dose (n=133,129,262) | 11.10 [9.39 to 13.13] | 8.25 [6.80 to 10.01] | 9.59 [8.44 to 10.90]
  Serotype 7F: After 13vPnC Dose 3 (n=133,130,263) | 5.05 [4.39 to 5.81] | 5.88 [4.93 to 7.02] | 5.44 [4.87 to 6.09]
  Serotype 7F: After 23vPS Dose (n=133,130,263) | 5.15 [4.50 to 5.90] | 5.93 [5.02 to 7.00] | 5.52 [4.96 to 6.14]
  Serotype 9V: After 13vPnC Dose 3 (n=133,130,263) | 5.02 [4.40 to 5.72] | 5.49 [4.59 to 6.57] | 5.25 [4.70 to 5.86]
  Serotype 9V: After 23vPS Dose (n=133,130,263) | 5.27 [4.62 to 6.00] | 5.83 [4.88 to 6.96] | 5.54 [4.96 to 6.18]
  Serotype 14: After 13vPnC Dose 3 (n=133,130,263) | 13.18 [10.19 to 17.05] | 15.35 [11.97 to 19.69] | 14.21 [11.89 to 16.98]
  Serotype 14: After 23vPS Dose (n=133,130,263) | 12.98 [10.10 to 16.67] | 16.24 [12.82 to 20.57] | 14.50 [12.21 to 17.21]
  Serotype 18C: After 13vPnC Dose 3 (n=132,130,262) | 3.84 [3.21 to 4.59] | 5.17 [4.25 to 6.28] | 4.45 [3.90 to 5.08]
  Serotype 18C: After 23vPS Dose (n=132,130,262) | 3.54 [2.98 to 4.20] | 4.80 [3.98 to 5.79] | 4.12 [3.62 to 4.68]
  Serotype 19A: After 13vPnC Dose 3 (n=133,130,263) | 14.16 [12.21 to 16.41] | 13.21 [11.13 to 15.68] | 13.68 [12.22 to 15.31]
  Serotype 19A: After 23vPS Dose (n=133,130,263) | 13.16 [11.31 to 15.33] | 13.28 [11.24 to 15.69] | 13.22 [11.82 to 14.79]
  Serotype 19F: After 13vPnC Dose 3 (n=130,127,257) | 6.15 [5.09 to 7.45] | 5.67 [4.47 to 7.19] | 5.91 [5.08 to 6.87]
  Serotype 19F: After 23vPS Dose (n=130,127,257) | 6.78 [5.65 to 8.14] | 5.84 [4.62 to 7.39] | 6.30 [5.44 to 7.30]
  Serotype 23F: After 13vPnC Dose 3 (n=132,129,261) | 6.69 [5.60 to 7.98] | 7.30 [5.87 to 9.09] | 6.98 [6.07 to 8.03]
  Serotype 23F: After 23vPS Dose (n=132,129,261) | 5.99 [5.05 to 7.11] | 7.03 [5.69 to 8.70] | 6.49 [5.66 to 7.43]

11. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody From 1 Month After 13vPnC Dose 3 to 1 Month After 23vPS Dose in Pediatric, Adult and All Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month after 13vPnC Dose 3 to 1 month after 23vPS Dose were computed using the logarithmically transformed assay results. Confidence interval (CI) for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both 1 month after 13vPnC Dose 3 and 1 month after 23vPS Dose blood draws.
Time Frame: 1 month after 13vPnC Dose 3, 1 month after 23vPS Dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 133 | 130 | 263
fold rise
  Serotype 1 (n = 128, 127, 255) | 1.08 [1.01 to 1.16] | 1.02 [0.96 to 1.08] | 1.05 [1.00 to 1.10]
  Serotype 3 (n = 124, 118, 242) | 1.11 [1.03 to 1.20] | 0.94 [0.88 to 1.00] | 1.02 [0.97 to 1.08]
  Serotype 4 (n = 133, 128, 261) | 1.00 [0.94 to 1.05] | 0.94 [0.90 to 0.99] | 0.97 [0.94 to 1.01]
  Serotype 5 (n = 132, 130, 262) | 1.07 [1.02 to 1.13] | 1.12 [1.05 to 1.19] | 1.09 [1.05 to 1.14]
  Serotype 6A (n = 122, 129, 251) | 0.97 [0.92 to 1.04] | 0.95 [0.91 to 0.99] | 0.96 [0.93 to 1.00]
  Serotype 6B (n = 133, 129, 262) | 0.91 [0.87 to 0.95] | 1.00 [0.96 to 1.04] | 0.95 [0.92 to 0.98]
  Serotype 7F (n = 133, 130, 263) | 1.02 [0.97 to 1.07] | 1.01 [0.95 to 1.06] | 1.01 [0.98 to 1.05]
  Serotype 9V (n = 133, 130, 263) | 1.05 [1.00 to 1.10] | 1.06 [1.01 to 1.11] | 1.06 [1.02 to 1.09]
  Serotype 14 (n = 133, 130, 263) | 0.98 [0.91 to 1.06] | 1.06 [0.99 to 1.13] | 1.02 [0.97 to 1.07]
  Serotype 18C (n = 132, 130, 262) | 0.92 [0.88 to 0.96] | 0.93 [0.89 to 0.97] | 0.92 [0.90 to 0.95]
  Serotype 19A (n = 133, 130, 263) | 0.93 [0.89 to 0.97] | 1.01 [0.96 to 1.05] | 0.97 [0.94 to 1.00]
  Serotype 19F (n = 130, 127, 257) | 1.10 [1.04 to 1.17] | 1.03 [0.97 to 1.09] | 1.07 [1.02 to 1.11]
  Serotype 23F (n = 132, 129, 261) | 0.90 [0.86 to 0.94] | 0.96 [0.91 to 1.02] | 0.93 [0.89 to 0.96]

12. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) 1 Month After 13vPnC Dose 3 and 1 Month After 23vPS Dose in Pediatric, Adult and All Participants
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of pediatric, adult and all participants using a mcOPA assay. GMT (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for both after 13vPnC Dose 3 and after 23vPS Dose blood draws. CI for GMT were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after 13vPnC Dose 3, 1 month after 23vPS Dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 132 | 128 | 260
titers
  Serotype 1: After 13vPnC Dose 3 (n=131,125,256) | 70 [53.4 to 93.0] | 67 [50.2 to 90.6] | 69 [56.4 to 84.3]
  Serotype 1: After 23vPS Dose (n=131,125,256) | 100 [76.6 to 130.3] | 66 [49.0 to 90.2] | 82 [66.9 to 100.2]
  Serotype 3: After 13vPnC Dose 3 (n=132,128,260) | 114 [94.6 to 136.7] | 78 [61.3 to 98.7] | 94 [81.1 to 109.7]
  Serotype 3: After 23vPS Dose (n=132,128,260) | 148 [123.9 to 177.3] | 103 [81.6 to 130.9] | 124 [107.0 to 144.0]
  Serotype 4: After 13vPnC Dose 3 (n=127,126,253) | 3213 [2698.5 to 3826.6] | 1888 [1427.3 to 2498.1] | 2466 [2087.0 to 2913.5]
  Serotype 4: After 23vPS Dose (n=127,126,253) | 3553 [2984.9 to 4229.7] | 1831 [1366.0 to 2453.7] | 2554 [2146.3 to 3038.7]
  Serotype 5: After 13vPnC Dose 3 (n=129,124,253) | 270 [197.0 to 370.1] | 143 [97.5 to 209.6] | 198 [154.2 to 253.5]
  Serotype 5: After 23vPS Dose (n=129,124,253) | 378 [276.5 to 516.9] | 186 [130.9 to 264.4] | 267 [210.6 to 338.6]
  Serotype 6A: After 13vPnC Dose 3 (n=132,127,259) | 8011 [6580.0 to 9752.1] | 2956 [2240.1 to 3900.3] | 4913 [4109.7 to 5873.6]
  Serotype 6A: After 23vPS Dose (n=132,127,259) | 7236 [5936.2 to 8819.4] | 2707 [2060.8 to 3556.3] | 4468 [3743.3 to 5333.1]
  Serotype 6B: After 13vPnC Dose 3 (n=130,126,256) | 7102 [5853.9 to 8615.8] | 3666 [2720.7 to 4940.5] | 5129 [4283.9 to 6141.0]
  Serotype 6B: After 23vPS Dose (n=130,126,256) | 6652 [5460.8 to 8102.8] | 3324 [2496.6 to 4426.2] | 4728 [3961.1 to 5643.2]
  Serotype 7F: After 13vPnC Dose 3 (n=131,125,256) | 4640 [3915.9 to 5497.9] | 2821 [2283.2 to 3484.4] | 3639 [3171.6 to 4174.8]
  Serotype 7F: After 23vPS Dose (n=131,125,256) | 5260 [4470.4 to 6189.9] | 3027 [2455.7 to 3731.3] | 4016 [3508.3 to 4597.9]
  Serotype 9V: After 13vPnC Dose 3 (n=127,125,252) | 4501 [3606.4 to 5618.0] | 1980 [1394.6 to 2811.7] | 2995 [2424.2 to 3700.8]
  Serotype 9V: After 23vPS Dose (n=127,125,252) | 5114 [4090.6 to 6393.0] | 2037 [1452.6 to 2857.6] | 3240 [2629.5 to 3991.2]
  Serotype 14: After 13vPnC Dose 3 (n=127,126,253) | 4023 [3317.5 to 4879.5] | 1431 [1115.7 to 1836.1] | 2405 [2030.8 to 2847.1]
  Serotype 14: After 23vPS Dose (n=127,126,253) | 4718 [3861.6 to 5764.9] | 1620 [1284.5 to 2043.0] | 2771 [2346.9 to 3270.7]
  Serotype 18C: After 13vPnC Dose 3 (n=129,121,250) | 5455 [4401.5 to 6761.4] | 1667 [1172.5 to 2370.8] | 3074 [2479.2 to 3810.5]
  Serotype 18C: After 23vPS Dose (n=129,121,250) | 6468 [5341.1 to 7832.2] | 1835 [1328.1 to 2535.5] | 3515 [2878.5 to 4292.8]
  Serotype 19A: After 13vPnC Dose 3 (n=131,125,256) | 1021 [837.5 to 1245.6] | 603 [456.7 to 796.3] | 790 [665.2 to 937.4]
  Serotype 19A: After 23vPS Dose (n=131,125,256) | 1244 [1012.1 to 1529.5] | 691 [531.0 to 898.6] | 933 [788.2 to 1105.5]
  Serotype 19F: After 13vPnC Dose 3 (n=126,117,243) | 1166 [884.3 to 1537.7] | 564 [375.0 to 848.1] | 822 [642.8 to 1051.0]
  Serotype 19F: After 23vPS Dose (n=126,117,243) | 1696 [1296.5 to 2217.5] | 790 [547.5 to 1139.7] | 1174 [934.2 to 1474.8]
  Serotype 23F: After 13vPnC Dose 3 (n=128,126,254) | 2346 [1883.3 to 2922.6] | 650 [435.3 to 969.9] | 1241 [976.6 to 1576.7]
  Serotype 23F: After 23vPS Dose (n=128,126,254) | 2595 [2143.3 to 3141.5] | 580 [386.1 to 871.8] | 1234 [970.1 to 1570.3]

13. Other Pre Specified Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From 1 Month After 13vPnC Dose 3 to 1 Month After 23vPS Dose in Pediatric, Adult and All Participants
Description: as for outcome 11
Time Frame: 1 month after 13vPnC Dose 3, 1 month after 23vPS Dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 132 | 128 | 260
fold rise
  Serotype 1 (n = 131, 125, 256) | 1.4 [1.23 to 1.63] | 1.0 [0.86 to 1.13] | 1.2 [1.08 to 1.31]
  Serotype 3 (n = 132, 128, 260) | 1.3 [1.15 to 1.48] | 1.3 [1.17 to 1.51] | 1.3 [1.20 to 1.44]
  Serotype 4 (n = 127, 126, 253) | 1.1 [1.04 to 1.18] | 1.0 [0.87 to 1.09] | 1.0 [0.97 to 1.10]
  Serotype 5 (n = 129, 124, 253) | 1.4 [1.15 to 1.71] | 1.3 [1.13 to 1.50] | 1.4 [1.20 to 1.53]
  Serotype 6A (n = 132, 127, 259) | 0.9 [0.85 to 0.96] | 0.9 [0.86 to 0.97] | 0.9 [0.87 to 0.95]
  Serotype 6B (n = 130, 126, 256) | 0.9 [0.87 to 1.01] | 0.9 [0.79 to 1.04] | 0.9 [0.86 to 0.99]
  Serotype 7F (n = 131, 125, 256) | 1.1 [1.06 to 1.21] | 1.1 [0.93 to 1.23] | 1.1 [1.02 to 1.19]
  Serotype 9V (n = 127, 125, 252) | 1.1 [1.05 to 1.23] | 1.0 [0.84 to 1.27] | 1.1 [0.97 to 1.21]
  Serotype 14 (n = 127, 126, 253) | 1.2 [1.07 to 1.28] | 1.1 [1.03 to 1.24] | 1.2 [1.08 to 1.23]
  Serotype 18C (n = 129, 121, 250) | 1.2 [1.04 to 1.35] | 1.1 [0.92 to 1.31] | 1.1 [1.03 to 1.27]
  Serotype 19A (n = 131, 125, 256) | 1.2 [1.11 to 1.34] | 1.1 [1.03 to 1.27] | 1.2 [1.10 to 1.27]
  Serotype 19F (n = 126, 117, 243) | 1.5 [1.25 to 1.69] | 1.4 [1.14 to 1.72] | 1.4 [1.26 to 1.62]
  Serotype 23F (n = 128, 126, 254) | 1.1 [0.96 to 1.28] | 0.9 [0.81 to 0.98] | 1.0 [0.91 to 1.09]

14. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-Specified Local Reactions: 13vPnC Dose 1
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling were scaled as Any (redness present or swelling present); Mild (0.5 to 2.0 centimeters (cm) for participants aged 6 to <12 years and 2.5 to 5.0 cm for participants aged greater than (>) 12 years); Moderate (2.5 to 7.0 cm for participants aged 6 to <12 years and 5.1 to 10.0 cm for participants aged >12 years); Severe (>7 cm for participants aged 6 to <12 years and >10 cm for participants aged >12 years). Pain at injection site was scaled as Any (pain present); Mild (did not interfere with activity); Moderate (interfered with activity); Severe (prevented daily activity). Report of severe swelling was confirmed as data entry error.
Time Frame: Within 14 days after 13vPnC Dose 1
Population: Safety population. Here "N" (number of participants analyzed) signifies participants with known values for any local reaction and "n" signifies participants with known values for specified local reaction. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 120 | 123 | 243
percentage of participants
  Redness: Any (n = 92, 88, 180) | 20.7 | 2.3 | 11.7
  Redness: Mild (n = 91, 88, 179) | 19.8 | 2.3 | 11.2
  Redness: Moderate (n = 85, 88, 173) | 2.4 | 0.0 | 1.2
  Redness: Severe (n = 84, 88, 172) | 0.0 | 0.0 | 0.0
  Swelling: Any (n = 97, 94, 191) | 29.9 | 9.6 | 19.9
  Swelling: Mild (n = 91, 93, 184) | 17.6 | 8.6 | 13.0
  Swelling: Moderate (n = 92, 89, 181) | 16.3 | 1.1 | 8.8
  Swelling: Severe (n = 84, 88, 172) | 1.2 | 0.0 | 0.6
  Pain at Injection Site: Any (n = 117, 121, 238) | 68.4 | 62.8 | 65.5
  Pain at Injection Site: Mild (n = 112, 116, 228) | 55.4 | 56.0 | 55.7
  Pain at Injection Site: Moderate (n = 94, 94, 188) | 28.7 | 18.1 | 23.4
  Pain at Injection Site: Severe (n = 86, 89, 175) | 8.1 | 2.2 | 5.1

15. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-Specified Local Reactions: 13vPnC Dose 2
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling were scaled as Any (redness present or swelling present); Mild (0.5 to 2.0 cm for participants aged 6 to <12 years and 2.5 to 5.0 cm for participants aged >12 years); Moderate (2.5 to 7.0 cm for participants aged 6 to <12 years and 5.1 to 10.0 cm for participants aged >12 years); Severe (>7 cm for participants aged 6 to <12 years and >10 cm for participants aged >12 years). Pain at injection site was scaled as Any (pain present); Mild (did not interfere with activity); Moderate (interfered with activity); Severe (prevented daily activity).
Time Frame: Within 14 days after 13vPnC Dose 2
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 120 | 119 | 239
percentage of participants
  Redness: Any (n = 101, 86, 187) | 13.9 | 2.3 | 8.6
  Redness: Mild (n = 100, 86, 186) | 10.0 | 2.3 | 6.5
  Redness: Moderate (n = 95, 85, 180) | 4.2 | 0.0 | 2.2
  Redness: Severe (n = 93, 85, 178) | 1.1 | 0.0 | 0.6
  Swelling: Any (n = 103, 88, 191) | 25.2 | 8.0 | 17.3
  Swelling: Mild (n = 102, 88, 190) | 18.6 | 8.0 | 13.7
  Swelling: Moderate (n = 99, 85, 184) | 12.1 | 0.0 | 6.5
  Swelling: Severe (n = 93, 85, 178) | 0.0 | 0.0 | 0.0
  Pain at Injection Site: Any (n = 117, 119, 236) | 60.7 | 79.8 | 70.3
  Pain at Injection Site: Mild (n = 110, 117, 227) | 49.1 | 72.6 | 61.2
  Pain at Injection Site: Moderate (n= 103, 96, 199) | 24.3 | 27.1 | 25.6
  Pain at Injection Site: Severe (n = 93, 86, 179) | 5.4 | 3.5 | 4.5

16. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-Specified Local Reactions: 13vPnC Dose 3
Description: as for outcome 15
Time Frame: Within 14 days after 13vPnC Dose 3
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 104 | 109 | 213
percentage of participants
  Redness: Any (n = 84, 70, 154) | 8.3 | 0.0 | 4.5
  Redness: Mild (n = 83, 70, 153) | 7.2 | 0.0 | 3.9
  Redness: Moderate (n = 82, 70, 152) | 2.4 | 0.0 | 1.3
  Redness: Severe (n = 80, 70, 150) | 0.0 | 0.0 | 0.0
  Swelling: Any (n = 89, 71, 160) | 18.0 | 4.2 | 11.9
  Swelling: Mild (n = 86, 71, 157) | 10.5 | 4.2 | 7.6
  Swelling: Moderate (n = 84, 70, 154) | 9.5 | 0.0 | 5.2
  Swelling: Severe (n = 80, 70, 150) | 0.0 | 0.0 | 0.0
  Pain at Injection Site: Any (n = 104, 109, 213) | 52.9 | 69.7 | 61.5
  Pain at Injection Site: Mild (n = 96, 105, 201) | 41.7 | 63.8 | 53.2
  Pain at Injection Site: Moderate (n = 89, 78, 167) | 19.1 | 24.4 | 21.6
  Pain at Injection Site: Severe (n = 83, 73, 156) | 4.8 | 5.5 | 5.1

17. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-Specified Systemic Events: 13vPnC Dose 1
Description: Specific systemic events (fever >=38 degrees Celsius[C], fatigue, headache, vomiting, diarrhea, muscle pain, joint pain and use of medication to treat pain/fever) were prompted for each day, and reported using an electronic diary. Fatigue, headache, muscle pain and joint pain were scaled as: Any (symptom present); Mild (did not interfere with activity); Moderate (some interference with activity); Severe (prevented routine daily activity). Vomiting was scaled as: Any (vomiting present); Mild (1-2 times in 24 hours); Moderate (>2 times in 24 hours); Severe (required intravenous hydration). Diarrhea was scaled as: Any (diarrhea present); Mild (2-3 loose stools in 24 hours); Moderate (4-5 loose stools 24 hours); Severe (>=6 loose stools in 24 hours). All reporting of fever >40 degrees C except 2 participants and all reporting of severe vomiting, after 13vPnC Dose 1, were confirmed as data entry errors.
Time Frame: Within 14 days after 13vPnC Dose 1
Population: Safety population. Here "N" (number of participants analyzed) signifies participants with known values for any systemic event and "n" signifies participants with known values for specified systemic event. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 128 | 138 | 266
percentage of participants
  Fever: >=38 degrees C (n= 94, 95, 189) | 19.1 | 17.9 | 18.5
  Fever: >=38, <38.5 degrees C (n = 87, 92, 179) | 8.0 | 8.7 | 8.4
  Fever: >=38.5, <39 degrees C (n = 85, 89, 174) | 2.4 | 3.4 | 2.9
  Fever: >=39, =<40 degrees C (n = 86, 88, 174) | 4.7 | 2.3 | 3.4
  Fever: >40 degrees C (n = 88, 93, 181) | 6.8 | 8.6 | 7.7
  Fatigue: Any (n = 111, 119, 230) | 47.7 | 58.8 | 53.5
  Fatigue: Mild (n = 105, 113, 218) | 33.3 | 51.3 | 42.7
  Fatigue: Moderate (n = 96, 99, 195) | 26.0 | 28.3 | 27.2
  Fatigue: Severe (n = 86, 92, 178) | 9.3 | 8.7 | 9.0
  Headache: Any (n = 107, 113, 220) | 39.3 | 61.1 | 50.5
  Headache: Mild (n = 100, 109, 209) | 33.0 | 57.8 | 45.9
  Headache: Moderate (n = 94, 97, 191) | 18.1 | 22.7 | 20.4
  Headache: Severe (n = 87, 89, 176) | 6.9 | 9.0 | 8.0
  Vomiting: Any (n = 89, 91, 180) | 18.0 | 7.7 | 12.8
  Vomiting: Mild (n = 89, 91, 180) | 14.6 | 7.7 | 11.1
  Vomiting: Moderate (n = 84, 88, 172) | 2.4 | 0.0 | 1.2
  Vomiting: Severe (n = 85, 88, 173) | 2.4 | 0.0 | 1.2
  Diarrhea: Any (n = 94, 105, 199) | 25.5 | 34.3 | 30.2
  Diarrhea: Mild (n = 92, 104, 196) | 19.6 | 29.8 | 25.0
  Diarrhea: Moderate (n = 86, 91, 177) | 8.1 | 7.7 | 7.9
  Diarrhea: Severe (n = 85, 88, 173) | 1.2 | 1.1 | 1.2
  Muscle Pain: Any (n = 108, 118, 226) | 48.1 | 62.7 | 55.8
  Muscle Pain: Mild (n = 103, 110, 213) | 36.9 | 56.4 | 46.9
  Muscle Pain: Moderate (n = 89, 98, 187) | 19.1 | 19.4 | 19.3
  Muscle Pain: Severe (n = 86, 91, 177) | 5.8 | 5.5 | 5.6
  Joint Pain: Any (n = 100, 105, 205) | 34.0 | 42.9 | 38.5
  Joint Pain: Mild (n = 98, 101, 199) | 26.5 | 36.6 | 31.7
  Joint Pain: Moderate (n = 89, 95, 184) | 12.4 | 17.9 | 15.2
  Joint Pain: Severe (n = 84, 91, 175) | 4.8 | 4.4 | 4.6
  Use of Medication to Treat Pain (n = 101, 96, 197) | 33.7 | 24.0 | 28.9
  Use of Medication to Treat Fever (n=112, 107, 219) | 44.6 | 39.3 | 42.0

18. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-Specified Systemic Events: 13vPnC Dose 2
Description: Specific systemic events (fever >=38 degrees Celsius[C], fatigue, headache, vomiting, diarrhea, muscle pain, joint pain and use of medication to treat pain/fever) were prompted for each day, and reported using an electronic diary. Fatigue, headache, muscle pain and joint pain were scaled as: Any (symptom present); Mild (did not interfere with activity); Moderate (some interference with activity); Severe (prevented routine daily activity). Vomiting was scaled as: Any (vomiting present); Mild (1-2 times in 24 hours); Moderate (>2 times in 24 hours); Severe (required intravenous hydration). Diarrhea was scaled as: Any (diarrhea present); Mild (2-3 loose stools in 24 hours); Moderate (4-5 loose stools 24 hours); Severe (>=6 loose stools in 24 hours). All reporting of fever >40 degrees C and all reporting of severe vomiting, after 13vPnC Dose 2, were confirmed as data entry errors.
Time Frame: Within 14 days after 13vPnC Dose 2
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 123 | 120 | 243
percentage of participants
  Fever: >=38 degrees C (n= 102, 88, 190) | 16.7 | 11.4 | 14.2
  Fever: >=38, <38.5 degrees C (n = 96, 87, 183) | 7.3 | 9.2 | 8.2
  Fever: >=38.5, <39 degrees C (n = 98, 85, 183) | 6.1 | 1.2 | 3.8
  Fever: >=39, =<40 degrees C (n = 97, 87, 184) | 7.2 | 3.4 | 5.4
  Fever: >40 degrees C (n = 95, 85, 180) | 1.1 | 1.2 | 1.1
  Fatigue: Any (n = 106, 105, 211) | 33.0 | 48.6 | 40.8
  Fatigue: Mild (n = 104, 103, 207) | 24.0 | 42.7 | 33.3
  Fatigue: Moderate (n = 96, 88, 184) | 10.4 | 21.6 | 15.8
  Fatigue: Severe (n = 95, 88, 183) | 7.4 | 5.7 | 6.6
  Headache: Any (n = 101, 106, 207) | 28.7 | 49.1 | 39.1
  Headache: Mild (n = 97, 102, 199) | 18.6 | 40.2 | 29.6
  Headache: Moderate (n = 97, 93, 190) | 13.4 | 28.0 | 20.5
  Headache: Severe (n = 94, 88, 182) | 2.1 | 3.4 | 2.7
  Vomiting: Any (n = 96, 89, 185) | 10.4 | 10.1 | 10.3
  Vomiting: Mild (n = 94, 89, 183) | 6.4 | 9.0 | 7.7
  Vomiting: Moderate (n = 94, 85, 179) | 3.2 | 1.2 | 2.2
  Vomiting: Severe (n = 94, 85, 179) | 3.2 | 0.0 | 1.7
  Diarrhea: Any (n = 95, 95, 190) | 10.5 | 26.3 | 18.4
  Diarrhea: Mild (n = 94, 93, 187) | 7.4 | 24.7 | 16.0
  Diarrhea: Moderate (n = 93, 87, 180) | 3.2 | 8.0 | 5.6
  Diarrhea: Severe (n = 94, 85, 179) | 4.3 | 1.2 | 2.8
  Muscle Pain: Any (n = 112, 104, 216) | 37.5 | 52.9 | 44.9
  Muscle Pain: Mild (n = 105, 103, 208) | 25.7 | 46.6 | 36.1
  Muscle Pain: Moderate (n = 100, 91, 191) | 15.0 | 20.9 | 17.8
  Muscle Pain: Severe (n = 95, 85, 180) | 5.3 | 2.4 | 3.9
  Joint Pain: Any (n = 106, 95, 201) | 26.4 | 34.7 | 30.3
  Joint Pain: Mild (n = 100, 93, 193) | 16.0 | 29.0 | 22.3
  Joint Pain: Moderate (n = 99, 89, 188) | 11.1 | 12.4 | 11.7
  Joint Pain: Severe (n = 94, 85, 179) | 4.3 | 2.4 | 3.4
  Use of Medication to Treat Pain (n = 100, 91, 191) | 20.0 | 17.6 | 18.8
  Use of Medication to Treat Fever (n=102, 96, 198) | 28.4 | 26.0 | 27.3

19. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-Specified Systemic Events: 13vPnC Dose 3
Description: Specific systemic events (fever >=38 degrees Celsius[C], fatigue, headache, vomiting, diarrhea, muscle pain, joint pain and use of medication to treat pain/fever) were prompted for each day, and reported using an electronic diary. Fatigue, headache, muscle pain and joint pain were scaled as: Any (symptom present); Mild (did not interfere with activity); Moderate (some interference with activity); Severe (prevented routine daily activity). Vomiting was scaled as: Any (vomiting present); Mild (1-2 times in 24 hours); Moderate (>2 times in 24 hours); Severe (required intravenous hydration). Diarrhea was scaled as: Any (diarrhea present); Mild (2-3 loose stools in 24 hours); Moderate (4-5 loose stools 24 hours); Severe (>=6 loose stools in 24 hours). All reporting of fever >40 degrees C except 1 participant and all reporting of severe vomiting, after 13vPnC Dose 3, were confirmed as data entry errors.
Time Frame: Within 14 days after 13vPnC Dose 3
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 106 | 113 | 219
percentage of participants
  Fever: >=38 degrees C (n= 85, 73, 158) | 10.6 | 11.0 | 10.8
  Fever: >=38, <38.5 degrees C (n = 82, 73, 155) | 6.1 | 5.5 | 5.8
  Fever: >=38.5, <39 degrees C (n = 81, 72, 153) | 2.5 | 5.6 | 3.9
  Fever: >=39, =<40 degrees C (n = 82, 70, 152) | 2.4 | 2.9 | 2.6
  Fever: >40 degrees C (n = 83, 70, 153) | 3.6 | 1.4 | 2.6
  Fatigue: Any (n = 92, 91, 183) | 25.0 | 47.3 | 36.1
  Fatigue: Mild (n = 89, 88, 177) | 20.2 | 39.8 | 29.9
  Fatigue: Moderate (n = 83, 80, 163) | 6.0 | 25.0 | 15.3
  Fatigue: Severe (n = 83, 73, 156) | 4.8 | 8.2 | 6.4
  Headache: Any (n = 88, 89, 177) | 18.2 | 46.1 | 32.2
  Headache: Mild (n = 84, 87, 171) | 10.7 | 41.4 | 26.3
  Headache: Moderate (n = 83, 77, 160) | 8.4 | 19.5 | 13.8
  Headache: Severe (n = 82, 72, 154) | 3.7 | 6.9 | 5.2
  Vomiting: Any (n = 85, 74, 159) | 8.2 | 9.5 | 8.8
  Vomiting: Mild (n = 84, 72, 156) | 7.1 | 5.6 | 6.4
  Vomiting: Moderate (n = 82, 73, 155) | 2.4 | 5.5 | 3.9
  Vomiting: Severe (n = 81, 72, 153) | 1.2 | 2.8 | 2.0
  Diarrhea: Any (n = 81, 81, 162) | 4.9 | 28.4 | 16.7
  Diarrhea: Mild (n = 81, 79, 160) | 4.9 | 25.3 | 15.0
  Diarrhea: Moderate (n = 80, 73, 153) | 1.3 | 6.8 | 3.9
  Diarrhea: Severe (n = 81, 73, 154) | 1.2 | 4.1 | 2.6
  Muscle Pain: Any (n = 99, 92, 191) | 37.4 | 47.8 | 42.4
  Muscle Pain: Mild (n = 93, 89, 182) | 25.8 | 37.1 | 31.3
  Muscle Pain: Moderate (n = 85, 78, 163) | 12.9 | 24.4 | 18.4
  Muscle Pain: Severe (n = 84, 72, 156) | 8.3 | 5.6 | 7.1
  Joint Pain: Any (n = 91, 83, 174) | 24.2 | 32.5 | 28.2
  Joint Pain: Mild (n = 88, 82, 170) | 15.9 | 28.0 | 21.8
  Joint Pain: Moderate (n = 82, 77, 159) | 7.3 | 15.6 | 11.3
  Joint Pain: Severe (n = 81, 71, 152) | 2.5 | 2.8 | 2.6
  Use of Medication to Treat Pain (n = 90, 79, 169) | 17.8 | 21.5 | 19.5
  Use of Medication to Treat Fever (n = 89, 75, 164) | 20.2 | 20.0 | 20.1

ADVERSE EVENTS:
Time Frame: Informed consent through 6-month follow-up after 13vPnC Dose 3. Local reactions and systemic events assessed within 14 days after: 13vPnC Dose 1 (Day 1); 13vPnC Dose 2 (28-42 days after 13vPnC Dose 1); and 13vPnC Dose 3 (28-42 days after 13vPnC Dose 2)
Description: Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may=serious for 1 subject and=non-serious for another subject or subject may have experienced both a serious and non-serious episode of same event. AEs/SAEs=non-systematic assessment; local reactions and systemic events=systematic assessment.
Groups:
- Prior 13vPnC Dose 1: Participants >=6 years of age (all participants) who received at least 1 of 3 doses of 0.5 mL of 13vPnC intramuscularly 1 month apart, followed by 1 dose of 0.5 mL of 23vPS intramuscularly 1 month after 13vPnC Dose 3 (23vPS Dose), assessed between signing of informed consent form and before 13vPnC Dose 1.
- 13vPnC Dose 1: Participants >=6 years of age (all participants) who received a single dose of 0.5 mL of 13vPnC intramuscularly on Day 1 (13vPnC Dose 1), assessed between 13vPnC Dose 1 and before 13vPnC Dose 2.
- 13vPnC Dose 2: Participants >=6 years of age (all participants) who received a single dose of 0.5 mL of 13vPnC intramuscularly 1 month after 13vPnC Dose 1 (13vPnC Dose 2), assessed between 13vPnC Dose 2 and before 13vPnC Dose 3.
- 13vPnC Dose 3: Participants >=6 years of age (all participants) who received a single dose of 0.5 mL of 13vPnC intramuscularly 1 month after 13vPnC Dose 2 (13vPnC Dose 3), assessed between 13vPnC Dose 3 and before 23vPS Dose.
- 23vPS Dose: Participants >=6 years of age (all participants) who received a single dose of 0.5 mL of 23vPS intramuscularly 1 month after 13vPnC Dose 3 (23vPS Dose), assessed between 23vPS Dose and before 23vPS Dose blood draw 1 month after 23vPS Dose.
- Follow-up: Participants >=6 years of age (all participants) who received 3 doses of 0.5 mL of 13vPnC intramuscularly 1 month apart, followed by 1 dose of 0.5 mL of 23vPS intramuscularly 1 month after 13vPnC Dose 3 (23vPS Dose), assessed from 23vPS blood draw to the 6-month follow-up telephone contact after 13vPnC Dose 3.
Arm/Group | Prior 13vPnC Dose 1 | 13vPnC Dose 1 | 13vPnC Dose 2 | 13vPnC Dose 3 | 23vPS Dose | Follow-up
Serious Adverse Events (participants affected / at risk) | 1/301 | 1/301 | 4/290 | 1/286 | 0/282 | 1/282
Other Adverse Events (participants affected / at risk) | 16/301 | 216/301 | 171/290 | 137/286 | 31/282 | 2/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior 13vPnC Dose 1 (N=301) | 13vPnC Dose 1 (N=301) | 13vPnC Dose 2 (N=290) | 13vPnC Dose 3 (N=286) | 23vPS Dose (N=282) | Follow-up (N=282)
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Prior 13vPnC Dose 1 (N=301) | 13vPnC Dose 1 (N=301) | 13vPnC Dose 2 (N=290) | 13vPnC Dose 3 (N=286) | 23vPS Dose (N=282) | Follow-up (N=282)
Conjunctivitis (Eye disorders) | 1 | 1 | 0 | 0/186 | 1 | 0/182
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0/186 | 0 | 1/182
Fatigue (General disorders) | 0 | 3 | 0 | 0/186 | 0 | 0/182
Pyrexia (General disorders) | 0 | 2 | 2 | 0/186 | 1 | 0/182
Influenza like illness (General disorders) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Injection site pain (General disorders) | 0 | 0 | 0 | 1/186 | 6 | 0/182
Injection site reaction (General disorders) | 0 | 0 | 0 | 0/186 | 2 | 0/182
Injection site swelling (General disorders) | 0 | 0 | 0 | 0/186 | 2 | 0/182
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 0/186 | 2 | 0/182
Influenza (Infections and infestations) | 0 | 5 | 1 | 8/186 | 3 | 1/182
Gastroenteritis (Infections and infestations) | 0 | 3 | 0 | 0/186 | 0 | 0/182
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 4 | 1/186 | 0 | 0/182
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 1/186 | 1 | 1/182
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0/186 | 0 | 0/182
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1/186 | 0 | 0/182
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1/186 | 0 | 0/182
Rhinitis (Infections and infestations) | 1 | 1 | 2 | 4/186 | 2 | 0/182
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Tinea capitis (Infections and infestations) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 2/186 | 0 | 0/182
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Viraemia (Infections and infestations) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Body tinea (Infections and infestations) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1/186 | 1 | 1/182
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 1/186 | 0 | 0/182
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Varicella (Infections and infestations) | 3 | 0 | 0 | 1/186 | 0 | 0/182
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0/186 | 0 | 1/182
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0/186 | 0 | 1/182
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2/186 | 1 | 0/182
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1/186 | 1 | 0/182
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0/186 | 0 | 1/182
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Headache (Nervous system disorders) | 0 | 3 | 1 | 1/186 | 2 | 0/182
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3 | 1/186 | 4 | 0/182
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2/186 | 0 | 0/182
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0/186 | 0 | 0/182
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1/186 | 0 | 0/182
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0/186 | 0 | 0/182
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2/186 | 0 | 0/182
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0/186 | 1 | 0/182
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0/186 | 0 | 0/182
Redness (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 21/180 | 16/187 | 7/154 | 0/0 | 0/0
Redness (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 20/179 | 12/186 | 6/153 | 0/0 | 0/0
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 2/173 | 4/180 | 2/152 | 0/0 | 0/0
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 0/172 | 1/178 | 0/150 | 0/0 | 0/0
Swelling (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 38/191 | 33/191 | 19/160 | 0/0 | 0/0
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 24/184 | 26/190 | 12/157 | 0/0 | 0/0
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 16/181 | 12/184 | 8/154 | 0/0 | 0/0
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 1/172 | 0/178 | 0/150 | 0/0 | 0/0
Pain at injection site (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 156/238 | 166/236 | 131/213 | 0/0 | 0/0
Pain at injection site (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 127/228 | 139/227 | 107/201 | 0/0 | 0/0
Pain at injection site (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 44/188 | 51/199 | 36/167 | 0/0 | 0/0
Pain at injection site (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 9/175 | 8/179 | 8/156 | 0/0 | 0/0
Fever (≥38°C) (General disorders) | 0/0 | 35/189 | 27/190 | 17/158 | 0/0 | 0/0
Fever (≥38°C but <38.5°C) (General disorders) | 0/0 | 15/179 | 15/183 | 9/155 | 0/0 | 0/0
Fever (≥38.5°C but <39°C) (General disorders) | 0/0 | 5/174 | 7/183 | 6/153 | 0/0 | 0/0
Fever (≥39°C but ≤40°C) (General disorders) | 0/0 | 6/174 | 10/184 | 4/152 | 0/0 | 0/0
Fever (>40°C) (General disorders) | 0/0 | 14/181 | 2/180 | 4/153 | 0/0 | 0/0 — All reporting of fever >40 degrees C except 2 participants in 13vPnC Dose 1 and 1 participant in 13vPnC Dose 3 were confirmed as data entry errors.
Fatigue (Any) (General disorders) | 0/0 | 123/230 | 86/211 | 66/183 | 0/0 | 0/0
Fatigue (Mild) (General disorders) | 0/0 | 93/218 | 69/207 | 53/177 | 0/0 | 0/0
Fatigue (Moderate) (General disorders) | 0/0 | 53/195 | 29/184 | 25/163 | 0/0 | 0/0
Fatigue (Severe) (General disorders) | 0/0 | 16/178 | 12/183 | 10/156 | 0/0 | 0/0
Headache (Any) (General disorders) | 0/0 | 111/220 | 81/207 | 57/177 | 0/0 | 0/0
Headache (Mild) (General disorders) | 0/0 | 96/209 | 59/199 | 45/171 | 0/0 | 0/0
Headache (Moderate) (General disorders) | 0/0 | 39/191 | 39/190 | 22/160 | 0/0 | 0/0
Headache (Severe) (General disorders) | 0/0 | 14/176 | 5/182 | 8/154 | 0/0 | 0/0
Vomiting (Any) (General disorders) | 0/0 | 23/180 | 19/185 | 14/159 | 0/0 | 0/0
Vomiting (Mild) (General disorders) | 0/0 | 20/180 | 14/183 | 10/156 | 0/0 | 0/0
Vomiting (Moderate) (General disorders) | 0/0 | 2/172 | 4/179 | 6/155 | 0/0 | 0/0
Vomiting (Severe) (General disorders) | 0/0 | 2/173 | 3/179 | 3/153 | 0/0 | 0/0 — All reporting of severe vomiting were confirmed as data entry errors.
Diarrhea (Any) (General disorders) | 0/0 | 60/199 | 35/190 | 27/162 | 0/0 | 0/0
Diarrhea (Mild) (General disorders) | 0/0 | 49/196 | 30/187 | 24/160 | 0/0 | 0/0
Diarrhea (Moderate) (General disorders) | 0/0 | 14/177 | 10/180 | 6/153 | 0/0 | 0/0
Diarrhea (Severe) (General disorders) | 0/0 | 2/173 | 5/179 | 4/154 | 0/0 | 0/0
Muscle pain (Any) (General disorders) | 0/0 | 126/226 | 97/216 | 81/191 | 0/0 | 0/0
Muscle pain (Mild) (General disorders) | 0/0 | 100/213 | 75/208 | 57/182 | 0/0 | 0/0
Muscle pain (Moderate) (General disorders) | 0/0 | 36/187 | 34/191 | 30/163 | 0/0 | 0/0
Muscle pain (Severe) (General disorders) | 0/0 | 10/177 | 7/180 | 11/156 | 0/0 | 0/0
Joint pain (Any) (General disorders) | 0/0 | 79/205 | 61/201 | 49/174 | 0/0 | 0/0
Joint pain (Mild) (General disorders) | 0/0 | 63/199 | 43/193 | 37/170 | 0/0 | 0/0
Joint pain (Moderate) (General disorders) | 0/0 | 28/184 | 22/188 | 18/159 | 0/0 | 0/0
Joint pain (Severe) (General disorders) | 0/0 | 8/175 | 6/179 | 4/152 | 0/0 | 0/0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.